CLINICAL TRIAL: NCT04690582
Title: Enhancing the Effectiveness of Cognitive Processing Therapy Among Suicidal Military Veterans With PTSD
Brief Title: Improving Treatment Outcomes for Suicidal Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Craig Bryan, Stress, Trauma, and Resilience (STAR) Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020H0431
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Suicidal Ideation; Suicide, Attempted; Ptsd
Keywords: crisis response plan; safety planning; safety plan
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (Active Comparator): Participants will receive cognitive processing therapy (CPT) for PTSD combined with a self-guided safety plan. As a recommended standard care practice with suicidal patients, the combination of CPT and safety plan represents treatment as usual. The safety plan will be assigned during the first therapy session.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT); Behavioral: Safety Planning Intervention (SPI)
- Crisis Response Plan (CPT+CRP) (Experimental): Participants will receive cognitive processing therapy (CPT) for PTSD combined with a collaborative crisis response plan (CRP). The CRP includes many of the same elements as the safety plan (i.e., warning signs, self-management strategies, sources of social support, crisis services), but is created collaboratively by the patient with active input of their clinician rather than being self-guided. The CRP also includes a section focused on the participant's reasons for living, an addition that has been shown to increase positive emotional states (e.g., hope, optimism) and lead to faster reductions in suicidal intent. The CRP will be collaboratively created during the first therapy session.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT); Behavioral: Crisis Response Plan (CRP); Behavioral: Narrative Assessment

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — Cognitive processing therapy (CPT) is a specific type of cognitive behavioral therapy that has been effective in reducing symptoms of PTSD that have developed after experiencing a variety of traumatic events including child abuse, combat, rape and natural disasters. CPT is generally delivered over 12 sessions and helps patients learn how to challenge and modify unhelpful beliefs related to the trauma. In so doing, the patient creates a new understanding and conceptualization of the traumatic event so that it reduces its ongoing negative effects on current life. This treatment is strongly recommended for the treatment of PTSD.
Behavioral: Crisis Response Plan (CRP) — The crisis response plan (CRP) is a collaborative, patient-centered intervention that is typically handwritten on an index cards and focuses on several key components: (1) warning signs, (2) self-regulatory strategies, (3) reasons for living, (4) sources of social support, and (5) professional and crisis services.
  Arms: Crisis Response Plan (CPT+CRP)
Behavioral: Safety Planning Intervention (SPI) — The safety planning intervention (SPI) is a suicide-focused intervention typically handwritten on a pre-printed form that includes the following sections: (1) warning signs, (2) internal coping strategies, (3) people and social settings that provide distraction, (4) people who can offer help, (5) professionals or agencies they can contact during a crisis, and (6) making the environment safe.
  Arms: Treatment As Usual
Behavioral: Narrative Assessment — The narrative assessment is a patient-centered assessment approach in which the clinician invites the patient to share "the story" of a recent crisis or period of intense emotional distress. Patients are asked to identify the thoughts, emotions, and physical sensations experienced in the time leading up to this crisis, as well as the contextual and environmental characteristics surrounding the crisis. Information obtained from the narrative assessment is then used to help formulate a crisis response plan.
  Arms: Crisis Response Plan (CPT+CRP)

SUMMARY:
The efficacy of cognitive processing therapy (CPT) for reducing the symptoms of posttraumatic stress disorder (PTSD) across populations including military personnel and veterans is well supported. CPT also contributes to significant and rapid reductions in suicide ideation among people diagnosed with PTSD, although available evidence suggests this effect decays over time. Studies also show that approximately 1 in 6 people who begin CPT without suicide ideation will subsequently report suicidal thoughts at some point during or soon after completing treatment. Research focused on improving CPT's effects on suicide risk is therefore warranted. The primary aim of this study is to determine if the integration of a crisis response plan (CRP)--an empirically-supported procedure for reducing suicide ideation and attempts--can lead to faster reductions in suicide ideation among acutely suicidal veterans receiving CPT and prevent the development of suicide ideation among veterans who begin CPT without suicide ideation.

DETAILED DESCRIPTION:
Cognitive behavioral treatments tend to be the most highly efficacious treatments for PTSD. Cognitive Processing Therapy (CPT) is one such treatment that has garnered a significant amount of empirical support, with a recent metaanalysis showing it was the most effective treatment for PTSD, typically yielding a 50% or larger reduction in PTSD symptoms from pre- to posttreatment. Redutions in PTSD symptoms are similar in magnitude when CPT is delivered in a virtual or telehealth format as compared to face-to-face delivery. Long-term follow-up studies conducted in nonmilitary samples also suggest the beneficial effects of CPT endure for up to 10 years posttreatment. Clinical improvement and recovery rates tend to be higher among patients who complete CPT compared to those that drop out of treatment early. Data also suggest that PTSD outcomes are moderated by session frequency, such that CPT sessions spaced closer together yield better effects than CPT sessions that are spaced further apart.

In addition to reducing PTSD symptoms, recent studies indicate CPT is also associated with significant short-term reduction in suicide ideation, potentially due to its effects on PTSD and depression symptom severity. In some studies, suicide ideation increased in severity again several months after the conclusion of therapy, however, suggesting a period of increased vulnerability for suicide. Enhancing CPT with procedures that have been shown to significantly reduce suicidal thoughts and behaviors could serve to further reduce suicide risk during and after treatment completion. One such procedure is the crisis response plan (CRP), a collaborative, patient-centered intervention that is typically handwritten on an index cards and focuses on several key components: (1) warning signs, (2) self-regulatory strategies, (3) reasons for living, (4) sources of social support, and (5) professional and crisis services. In a randomized clinical trial previously conducted by our team, acutely suicidal patients who received a CRP showed significantly faster declines in suicide ideation and were 76% less likely to attempt suicide during the 6-month follow-up as compared to patients who received mental health treatment as usual.

In the present study, the investigators aim to determine if the addition of a CRP with CPT will lead to faster reductions in suicide ideation and prevent the recurrence of suicide ideation during follow-up as compared to the standard provision of CPT. To achieve this, this study includes a two-arm, double blind parallel randomized clinical trial. The investigators will enroll 150 military personnel and veterans who meet full diagnostic criteria for PTSD (i.e., having 4 of 4 symptom criteria at or above threshold levels) or subthreshold PTSD (i.e., having 3 of 4 symptom criteria at or above threshold levels). All participants will receive 10-12 sessions of CPT, administered on a daily basis for two consecutive weeks. The investigators will assess suicide ideation, suicide attempts, and psychological symptom severity for up to one year post-treatment. Our primary hypothesis is that the combination of CRP and CPT will result in larger reductions in suicide ideation than CPT alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Current or prior service in the U.S. military
* Current diagnosis of PTSD or subthreshold PTSD
* Ability to speak and understand the English language
* Ability to complete the informed consent process.

Exclusion Criteria:

* Substance use disorder requiring medical management
* Imminent suicide risk warranting inpatient hospitalization or suicide-focused treatment
* Impaired mental status that precludes the ability to provide informed consent (e.g., intoxication, psychosis, mania)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Bryan, PsyD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in using IPD and/or computer code collected or generated as part of this study may do so by contacting the study PI. Researchers will be asked to complete a Data Use Request Form, which includes contact information, description of the research project for which the data and/or code would be used, specification of which data and/or code would be needed for their proposed project, an approximate time line for their proposed project, and authorship on their proposed project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of primary results
Access Criteria: All requests for data and/or code use will be reviewed by the PIs and co-Is and a majority vote will be used to determine whether the request is approved or not. If the request is approved, Dr. Bryan will inform the requestor, return a signed copy of the completed Data Use Request Form to the requestor, and let the requestor know that written IRB approval of the requestor's proposed study from the requestor's home institution will be required before data and/or code will be shared with the requestor. If a request is approved pending revision to the Data Use Request Form, Dr. Bryan will work with requestors to revise sections of their Data Use Request Forms in order to obtain approval. If the request is not approved, Dr. Bryan will inform the requestor and returned a signed copy of the completed Data Use Request Form to the requestor that includes an explanation for the denial.

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Plan: Participants will receive cognitive processing therapy (CPT) for PTSD combined with a self-guided safety plan. As a recommended standard care practice with suicidal patients, the combination of CPT and safety plan represents treatment as usual. The safety plan will be assigned during the first therapy session.
  Safety Plan (SP): Safety planning (SP) is a suicide-focused intervention typically handwritten on a pre-printed form that includes the following sections: (1) warning signs, (2) internal coping strategies, (3) people and social settings that provide distraction, (4) people who can offer help, (5) professionals or agencies they can contact during a crisis, and (6) making the environment safe.
- Crisis Response Plan: Participants will receive cognitive processing therapy (CPT) for PTSD combined with a collaborative crisis response plan (CRP). The CRP includes many of the same elements as the safety plan (i.e., warning signs, self-management strategies, sources of social support, crisis services), but is created collaboratively by the patient with active input of their clinician rather than being self-guided. The CRP begins with a narrative suicide risk assessment, in which the patient is invited to "tell the story" of their suicidal thoughts and/or behaviors. The CRP also includes a section focused on the participant's reasons for living, an addition that has been shown to increase positive emotional states (e.g., hope, optimism) and lead to faster reductions in suicidal intent. The CRP will be collaboratively created during the first therapy session.
  Crisis Response Plan (CRP): The crisis response plan (CRP) is a collaborative, patient-centered intervention that is typically handwritten on an index cards and focuses on several key components: (1) warning signs, (2) self-regulatory strategies, (3) reasons for living, (4) sources of social support, and (5) professional and crisis services.
Period: Overall Study
Arm/Group | Safety Plan | Crisis Response Plan
Started | 81 | 76
Completed | 75 | 72
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Plan | Crisis Response Plan | Total
Number analyzed (Participants) | 81 | 76 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 66 | 142
  >=65 years | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.0) | 48.3 (12.1) | 47.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 12 | 42
  Male | 51 | 64 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 63 | 58 | 121
  Black | 9 | 7 | 16
  Native American | 3 | 2 | 5
  Asian | 2 | 2 | 4
  Other | 4 | 7 | 11
  Latino/Hispanic | 3 | 10 | 13
Region of Enrollment [Number; unit: participants]
  United States | 81 | 76 | 157
Scale for Suicide Ideation [Mean (Standard Deviation); unit: units on a scale] — The Scale for Suicide Ideation is a self-report scale that assesses the intensity of suicide-related thoughts, urges, intentions, and behaviors. Scores range from 0 to 38, with higher scores indicating more severe suicide ideation.
  units on a scale | 5.91 (7.79) | 6.86 (7.56) | 6.37 (7.67)
Number of Participants with Pre-Baseline Suicide Attempts [Count of Participants; unit: Participants] — Pre-baseline suicide attempts was assessed with the Self-Injurious Thoughts and Behaviors Interview-Revised, a self-report scale that assesses a range of self-injurious behaviors including suicide attempts, interrupted suicide attempts, preparatory behaviors, and non-suicidal self-injury. Suicidal behaviors are coded with a binary variable indicating the presence or absence of any suicidal behavior during the study period.
  Participants | 62 | 63 | 125
National Stressful Events Survey PTSD Short Scale [Mean (Standard Deviation); unit: units on a scale] — The National Stressful Events Survey PTSD Short Scale is a 9-item self-report scale that assesses severity of PTSD symptoms. Scores range from 0 to 36, with higher scores indicating more severe PTSD symptoms.
  units on a scale | 27.01 (7.09) | 25.93 (7.38) | 26.49 (7.23)

OUTCOME MEASURES:

1. Primary Outcome: Change in Suicide Ideation
Description: Suicide ideation will be measured using the Scale for Suicide Ideation, an empirically-supported self-report scale that assesses the intensity of suicide-related thoughts, urges, intentions, and behaviors. Scores range from 0 to 38, with higher scores indicating more severe suicide ideation.
Time Frame: Baseline (Pretreatment), 1 week, 2 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Safety Plan | Crisis Response Plan
Number analyzed (Participants) | 81 | 76
units on a scale
  Baseline (Pretreatment) | 5.91 (7.79) | 6.37 (7.67)
  1 week | 3.67 (5.64) | 2.47 (4.83)
  2 weeks | 3.00 (5.49) | 2.25 (5.18)
  26 weeks | 3.49 (6.59) | 3.20 (6.22)
  52 weeks | 3.42 (5.32) | 3.36 (5.37)

2. Primary Outcome: Percent With Follow-up Suicidal Behaviors
Description: Percent of participants with one or more suicidal behaviors will be measured using the Self-Injurious Thoughts and Behaviors Interview-Revised, an empirically-supported self-report scale that assesses a range of self-injurious behaviors including suicide attempts, interrupted suicide attempts, preparatory behaviors, and non-suicidal self-injury during the 52 week follow-up. Suicidal behaviors will be coded with a binary variable indicating the presence or absence of any suicidal behavior during the study period.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Plan | Crisis Response Plan
Number analyzed (Participants) | 81 | 76
Participants | 4 | 3

3. Primary Outcome: Number of Follow-up Suicidal Behaviors
Description: Number of suicidal behaviors will be measured using the Self-Injurious Thoughts and Behaviors Interview-Revised, an empirically-supported self-report scale that assesses a range of self-injurious behaviors including suicide attempts, interrupted suicide attempts, preparatory behaviors, and non-suicidal self-injury during the 52 week follow-up. Suicidal behaviors will be coded with a binary variable indicating the presence or absence of any suicidal behavior during the study period and then summed to calculate the total number of suicidal behaviors during the 52 week follow-up.
Time Frame: 52 weeks
Measure: Number; unit: count of suicide attempts
Arm/Group | Safety Plan | Crisis Response Plan
Number analyzed (Participants) | 81 | 76
count of suicide attempts | 8 | 4

4. Secondary Outcome: Change in PTSD Symptoms
Description: Change in PTSD symptom severity will be measured using the National Stressful Events Survey PTSD Short Scale. Scores range from 0 to 36, with higher scores indicating more severe PTSD symptoms.
Time Frame: Baseline (Pretreatment) , 1 week, 2 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Safety Plan | Crisis Response Plan
Number analyzed (Participants) | 81 | 76
units on a scale
  Baseline (Pretreatment) | 27.01 (7.09) | 25.93 (7.38)
  1 week | 17.57 (7.59) | 18.05 (8.74)
  2 weeks | 13.42 (8.10) | 13.06 (6.85)
  26 weeks | 14.09 (9.22) | 14.87 (9.33)
  52 weeks | 14.85 (8.91) | 14.83 (9.44)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Safety Plan | Crisis Response Plan
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/76
Other Adverse Events (participants affected / at risk) | 0/81 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT04690582/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT04690582/ICF_001.pdf